CLINICAL TRIAL: NCT02247089
Title: The Effect of Massage Therapy to Control Night Shift Related Stress: A Pilot Prospective Randomized Crossover Trial
Brief Title: The Effect of Massage Therapy to Control Night Shift Related Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Registered Massage Therapists Association of British Columbia (Other)
Responsible Party: Principal Investigator, Mir Sohail Fazeli, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H13-01584
Record Dates: First submitted 2014-09-10; First posted 2014-09-23 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Stress
Keywords: Night Shift work; Stress; Autonomic nervous system (ANS); Heart rate variability (HRV); Pre-ejection period (PEP); Inflammation; Pro-inflammatory cytokines; Massage Therapy
MeSH Terms: conditions — Inflammation | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Massage Therapy — Intervention consists of administering a 30-minute-long upper body massage by a registered massage therapist following a massage protocol developed by Vancouver College of Massage Therapy (VCMT).
Other: Journal reading (No massage therapy) — Intervention consists of journal reading in the same sitting position as the massage therapy session for approximately 30 minutes.

SUMMARY:
Background:

The sympathetic and parasympathetic branches (SNS and PNS) of the autonomic nervous system (ANS), keep our body in a state of balance, which can be disturbed in situations of uncontrolled stress. Sleep deprivation and specifically night shift is a source of stress with adverse consequences on sleep, wakefulness, eating patterns and cardio-vascular function. Furthermore, imbalanced autonomic profile is also associated with increased inflammation, a known risk factor for cardiac problems, diabetes, and cancer.

Parasympathetic stimulation can control the inflammatory reaction, leading research toward interventions which can stimulate the cholinergic pathway. Among these interventions, massage therapy has shown to stimulate the PNS and bring back the balance within the body's organs.

Objectives:

1. To assess the physiological effects of night shifts on the ANS profile and bio-markers of inflammation and stress in blood
2. To assess whether one session of massage therapy can revert the adverse effects of night shift via re-balancing these components.

Methods:

A pilot prospective randomized crossover trial with 10 healthy hospital staff is in progress:

Each participants will be their own control. All participants will be measured for their baseline characteristics and outcomes of interest on a regular working day as well as at the end of 2 nights of shift work. At the end of one shift they will be randomly assigned to receive a 30-minute-long "upper body massage", while at the end of the other shift they will receive a "reading intervention" which would serve as a control intervention. Randomization is done using a computer system that also verifies inclusion-exclusion criteria before allocating the intervention.

The autonomic profile is measured by spectral analysis of Heart Rate Variability (HRV) captured by a state-of-the-art machine which non-invasively records electrical signals from the body. The inflammatory markers in the blood are also measured using top-notch laboratory technology.

The results of the study will be reported by comparing the outcomes of each subject with their own baseline as well as comparing the two interventions for the effect of massage. Data will be pooled for all subjects in order to show the overall effect.

The final results of this study will be used to plan stress management intervention trials.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy hospital staff between the ages of 20 to 60 taking rotating night shifts on a regular basis.

Exclusion Criteria:

* Participants who are on anti-depressants or drugs that affect the cardiovascular system or the ANS.
* Any conditions or disorders that would affect the cardiovascular system or the activity of the ANS.
* Participants who smoke more than 10 cigarettes/day.
* Inability to provide consent.
* Inability to speak and/or understand English.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) parameters | up to 1 month
  Main HRV parameters that will be reported include High Frequency (HF) which is the power in high frequency range representative of the parasympathetic nervous system activity, HFnu which is the HF power in normalized units, and total power which is the total variability of the autonomic nervous system over the temporal segment.
  The HRV parameters will be measured at 5 different time points all at approximately the same time in the morning. These 5 time points are as follows:
  1. Baseline measurement: This measurement takes place on a regular working day with no night shift at the end of the day or the night before.
  2. Shift measurements (Pre-intervention): These consist of measurements before interventions at the end of two separate nights of shift work.
  3. Post-intervention measurements: These consist of measurements after interventions at the end of two separate nights of shift work.
Pre-ejection period (PEP) | up to 1 month
  PEP is the time interval between electrical stimulation of the sinoatrial node and opening of the aortic valves and has shown to be inversely correlated with the activity of the sympathetic nervous system.
  PEP will be measured at 5 different time points all at approximately the same time in the morning. These 5 time points are as follows:
  1. Baseline measurement: This measurement takes place on a regular working day with no night shift at the end of the day or the night before.
  2. Shift measurements (Pre-intervention): These consist of measurements before interventions at the end of two separate nights of shift work.
  3. Post-intervention measurements: These consist of measurements after interventions at the end of two separate nights of shift work.

SECONDARY OUTCOMES:
Pro-inflammatory cytokines | 5 times within 1 month
  These consist of protein and mRNA levels of secreted pro-inflammatory cytokines (IL-6, IL-1beta and TNF-alpha) in blood.
  The pro-inflammatory cytokines will be measured at 5 different time points all at approximately the same time in the morning. These 5 time points are as follows:
  1. Baseline measurement: This measurement takes place on a regular working day with no night shift at the end of the day or the night before.
  2. Shift measurements (Pre-intervention): These consist of measurements before interventions at the end of two separate nights of shift work.
  3. Post-intervention measurements: These consist of measurements after interventions at the end of two separate nights of shift work.
Plasma Cortisol level | 5 times within 1 month
  The plasma cortisol level will be measured at 5 different time points all at approximately the same time in the morning. These 5 time points are as follows:
  1. Baseline measurement: This measurement takes place on a regular working day with no night shift at the end of the day or the night before.
  2. Shift measurements (Pre-intervention): These consist of measurements before interventions at the end of two separate nights of shift work.
  3. Post-intervention measurements: These consist of measurements after interventions at the end of two separate nights of shift work.

OTHER OUTCOMES:
Blood Pressure | 5 times within 1 month
  Systolic and diastolic Blood pressure will be measure at 5 different time points all at approximately the same time in the morning. These 5 time points are as follows:
  1. Baseline measurement: This measurement takes place on a regular working day with no night shift at the end of the day or the night before.
  2. Shift measurements (Pre-intervention): These consist of measurements before interventions at the end of two separate nights of shift work.
  3. Post-intervention measurements: These consist of measurements after interventions at the end of two separate nights of shift work.
Heart Rate | 5 times within 1 month
  Average of beat to beat heart rate (in beats per minute) will be measured at 5 different time points all at approximately the same time in the morning. These 5 time points are as follows:
  1. Baseline measurement: This measurement takes place on a regular working day with no night shift at the end of the day or the night before.
  2. Shift measurements (Pre-intervention): These consist of measurements before interventions at the end of two separate nights of shift work.
  3. Post-intervention measurements: These consist of measurements after interventions at the end of two separate nights of shift work.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Collet, MD, PhD, Principal Investigator — Children's & Women's Health Centre of British Columbia; Mir Sohail Fazeli, MD, PhD Candidate, Principal Investigator — The University of British Columbia
Locations (1):
- BC Children's and Women's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Fazeli MS, Pourrahmat MM, Massah G, Lee K, Lavoie PM, Fazeli M, Esser A, Collet JP. The Effect of Massage on the Cardiac Autonomic Nervous System and Markers of Inflammation in Night Shift Workers: a Pilot Randomized Crossover Trial. Int J Ther Massage Bodywork. 2020 Aug 27;13(3):6-17. eCollection 2020 Sep. PMID 32922577